CLINICAL TRIAL: NCT01076205
Title: Long Term Documentation of the Safety and Efficacy as Well as the Effects on Quality of Life and Work Productivity in Patients With Rheumatoid Arthritis Under HUMIRA® (Adalimumab) in Routine Clinical Practice (AGIL)
Brief Title: Safety and Effect on Quality of Life/Work Productivity of Humira in Patients With Rheumatoid Arthritis
Acronym: AGIL
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-973
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Work Productivity; Long-term Observation; Humira; Quality of Life; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Adults with moderate to severe active rheumatoid arthritis (RA) who initiated adalimumab therapy during routine clinical care.

SUMMARY:
The AGIL study was designed to evaluate the effectiveness and safety of adalimumab over 5 years in routine daily clinical practice in Germany, with a focus on the impact of therapy on employment-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active rheumatoid arthritis in adults with insufficient response to disease-modifying antirheumatic drugs
* Inclusive methotrexate
* Moderate to severe active rheumatoid arthritis in adults who have not been treated with methotrexate before; In case of incompatibility with methotrexate, Humira can be used as monotherapy.

Exclusion Criteria:

* Hypersensitivity against the drug or one of the other ingredients
* Active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections)
* Moderate to severe cardiac insufficiency

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample: Patients with rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 7229 (Actual)
Dates: Start 2009-01-12 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kleine, PhD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- [Derived] Behrens F, Tony HP, Koehm M, Schwaneck EC, Gnann H, Greger G, Burkhardt H, Schmalzing M. Sustained improvement in work outcomes in employed patients with rheumatoid arthritis during 2 years of adalimumab therapy: an observational cohort study. Clin Rheumatol. 2020 Sep;39(9):2583-2592. doi: 10.1007/s10067-020-05038-y. Epub 2020 Mar 23. PMID 32206973
- [Derived] Behrens F, Koehm M, Schwaneck EC, Schmalzing M, Gnann H, Greger G, Tony HP, Burkhardt H. Use of a "critical difference" statistical criterion improves the predictive utility of the Health Assessment Questionnaire-Disability Index score in patients with rheumatoid arthritis. BMC Rheumatol. 2019 Dec 10;3:51. doi: 10.1186/s41927-019-0095-2. eCollection 2019. PMID 31867564
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with rheumatoid arthritis (RA) were enrolled at 326 clinical centers in Germany and seen during regular visits for routine clinical care.
Groups:
- Adalimumab: Participants with moderate to severe active rheumatoid arthritis who initiated adalimumab therapy during routine clinical care.
Period: Overall Study
Arm/Group | Adalimumab
Started | 7229
Completed (Participants who were ongoing at the 60 month visit.) | 1210
Not Completed | 6019
Not completed — Adverse Drug Reaction | 299
Not completed — Lack of Effectiveness | 1423
Not completed — Other Reason | 1075
Not completed — Unknown Reason | 71
Not completed — Lost to Follow-up | 3151

BASELINE CHARACTERISTICS:
Population: The safety set included all enrolled participants who received at least one dose of adalimumab.
Arm/Group | Adalimumab
Number analyzed (Participants) | 7229
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 7165
    (all) | 54.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants with available data
  Participants
    number analyzed (Participants) | 7176
    Female | 5267
    Male | 1909
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Disease [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 7039
    (all) | 9.6 (8.8)
Number of Missed Work Days in Last 6 Months [Mean (Standard Deviation); unit: days] — Population: Participants who were employed part-time or full-time
  days
    number analyzed (Participants) | 3887
    (all) | 19.9 (41.7)
Work Productivity and Activity Impairment [Mean (Standard Deviation); unit: percent impairment] — The Work Productivity and Activity Impairment (WPAI) questionnaire for general health is a validated tool in RA consisting of 6 questions, based on patient recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), total work productivity impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health. WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes. Population: Participants with available WPAI data; The first 3 scores were assessed in participants who were employed.
  percent impairment
    Absenteeism: number analyzed (Participants) | 2362
    Absenteeism | 21.4 (36.9)
    Presenteeism: number analyzed (Participants) | 3046
    Presenteeism | 47.2 (27.3)
    Total work productivity impairment: number analyzed (Participants) | 2124
    Total work productivity impairment | 50.9 (29.2)
    Total activity impairment: number analyzed (Participants) | 6862
    Total activity impairment | 54.9 (25.0)
Work Activity Index [Mean (Standard Deviation); unit: units on a scale] — The WAI is a tool designed to record the work ability of employees and consists of 7 questions. The modified WAI used in this study included Questions 1, 2, 4, 6, and 7 of the WAI. Question 3, which involves the number of current diseases diagnosed by a physician, was omitted because this parameter was unlikely to reflect change due to treatment. Question 5 (sick leave during the past year) was replaced with the previous question concerning sick leave days. WAI scores range from 7 (worst) to 49 (best). Population: Participants who were employed part-time or full-time
  units on a scale
    number analyzed (Participants) | 2183
    (all) | 32.1 (7.8)
Disease Activity Score - 28 Joints (DAS28) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score < 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 6132
    (all) | 4.63 (1.51)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. Population: Participants with available data
  joints
    number analyzed (Participants) | 7111
    (all) | 7.4 (6.8)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. Population: Participants with available data
  joints
    number analyzed (Participants) | 7111
    (all) | 5.0 (5.3)
Erythrocyte Sedimentation Rate [Mean (Standard Deviation); unit: mm/hr] — Population: Participants with available data
  mm/hr
    number analyzed (Participants) | 6348
    (all) | 26.5 (21.7)
C-reactive Protein [Mean (Standard Deviation); unit: mg/L] — Population: Participants with available data
  mg/L
    number analyzed (Participants) | 6764
    (all) | 17.3 (48.7)
Health-Assessment Questionnaire-Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing, eating, walking, and hygiene. Patients are asked about their ability to complete these tasks in the past week on the following scale: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 6977
    (all) | 1.19 (0.74)
Euroqol Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — EuroQol-5 Dimensions (EQ-5D) is a generic instrument for measuring health-related quality of life. The VAS is a vertical scale ranging from 0 to 100 that provides a patient-reported assessment of overall health. Patients are asked to mark how good or bad their health is on that day, with 100 meaning "the best health you can imagine" and 0 meaning "the worst health you can imagine." Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 6912
    (all) | 52.2 (22.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Missed Working Days Due to Sick Leave in the Past 6 Months
Description: Primary effectiveness outcomes related to employment were performed in patients who were employed part- or full-time at baseline. Sick leave days were based on patient recall.
Time Frame: Baseline and 6, 12, 24, 36, 48, and 60 months
Population: Participants who were employed outside of the home, on either a part-time or full-time basis, at baseline (employed patient set), with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adalimumab
Number analyzed (Participants) | 3156
days
  Month 6: number analyzed (Participants) | 2267
  Month 6 | -4.3 (32.7)
  Month 12: number analyzed (Participants) | 1855
  Month 12 | -3.4 (37.3)
  Month 24: number analyzed (Participants) | 1290
  Month 24 | -5.6 (30.3)
  Month 36: number analyzed (Participants) | 868
  Month 36 | -6.7 (32.2)
  Month 48: number analyzed (Participants) | 596
  Month 48 | -6.4 (27.7)
  Month 60: number analyzed (Participants) | 415
  Month 60 | -4.1 (32.0)

2. Primary Outcome: Percentage of Participants With > 5 Missed Working Days Due to Sick Leave in the Past 6 Months
Description: as for outcome 1
Time Frame: Baseline, 6, 12, 24, 36, 48, and 60 months
Population: Participants who were employed outside of the home, on either a part-time or full-time basis, at baseline (employed patient set), with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 3156
percentage of participants
  Baseline | 44.7
  Month 6: number analyzed (Participants) | 2326
  Month 6 | 29.5
  Month 12: number analyzed (Participants) | 1906
  Month 12 | 28.5
  Month 24: number analyzed (Participants) | 1321
  Month 24 | 27.9
  Month 36: number analyzed (Participants) | 890
  Month 36 | 26.2
  Month 48: number analyzed (Participants) | 613
  Month 48 | 24.1
  Month 60: number analyzed (Participants) | 426
  Month 60 | 26.1

3. Primary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Absenteeism
Description: The Work Productivity and Activity Impairment (WPAI) questionnaire for general health is a validated tool in RA consisting of 6 questions, based on patient recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), total work productivity impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health.
  WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes.
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: Participants who were employed outside of the home, on either a part-time or full-time basis, at baseline (employed patient set) and at each time point, and with available WPAI data.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 2253
percent impairment
  Month 3: number analyzed (Participants) | 1482
  Month 3 | -7.9 (34.6)
  Month 6: number analyzed (Participants) | 1220
  Month 6 | -8.0 (37.2)
  Month 12: number analyzed (Participants) | 969
  Month 12 | -7.3 (38.3)
  Month 24: number analyzed (Participants) | 660
  Month 24 | -6.5 (36.1)
  Month 36: number analyzed (Participants) | 424
  Month 36 | -8.0 (34.7)
  Month 48: number analyzed (Participants) | 287
  Month 48 | -5.2 (34.6)
  Month 60: number analyzed (Participants) | 200
  Month 60 | -5.2 (40.7)

4. Primary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Presenteeism
Description: as for outcome 3
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 2758
percent impairment
  Month 3: number analyzed (Participants) | 2157
  Month 3 | -11.3 (25.8)
  Month 6: number analyzed (Participants) | 1852
  Month 6 | -11.8 (26.7)
  Month 12: number analyzed (Participants) | 1513
  Month 12 | -12.7 (28.2)
  Month 24: number analyzed (Participants) | 1084
  Month 24 | -12.9 (28.6)
  Month 36: number analyzed (Participants) | 717
  Month 36 | -15.3 (28.8)
  Month 48: number analyzed (Participants) | 490
  Month 48 | -16.4 (29.4)
  Month 60: number analyzed (Participants) | 343
  Month 60 | -15.2 (27.8)

5. Primary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Total Work Productivity Impairment
Description: as for outcome 3
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 2026
percent impairment
  Month 3: number analyzed (Participants) | 1313
  Month 3 | -13.0 (27.7)
  Month 6: number analyzed (Participants) | 1073
  Month 6 | -14.4 (28.8)
  Month 12: number analyzed (Participants) | 851
  Month 12 | -16.4 (30.3)
  Month 24: number analyzed (Participants) | 596
  Month 24 | -15.3 (30.6)
  Month 36: number analyzed (Participants) | 382
  Month 36 | -18.8 (29.3)
  Month 48: number analyzed (Participants) | 261
  Month 48 | -16.7 (31.6)
  Month 60: number analyzed (Participants) | 171
  Month 60 | -16.5 (33.8)

6. Primary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Total Activity Impairment
Description: as for outcome 3
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: Participants who were employed outside of the home, on either a part-time or full-time basis, at baseline (employed patient set) and with available WPAI data.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 3248
percent impairment
  Month 3: number analyzed (Participants) | 2758
  Month 3 | -11.9 (26.5)
  Month 6: number analyzed (Participants) | 2420
  Month 6 | -12.8 (27.5)
  Month 12: number analyzed (Participants) | 2007
  Month 12 | -13.8 (28.6)
  Month 24: number analyzed (Participants) | 1424
  Month 24 | -14.3 (28.4)
  Month 36: number analyzed (Participants) | 970
  Month 36 | -15.4 (29.7)
  Month 48: number analyzed (Participants) | 687
  Month 48 | -14.8 (29.4)
  Month 60: number analyzed (Participants) | 509
  Month 60 | -14.8 (28.6)

7. Primary Outcome: Change From Baseline in Work Activity Index (WAI)
Description: The WAI is a tool designed to record the work ability of employees and consists of 7 questions. The modified WAI used in this study included Questions 1, 2, 4, 6, and 7 of the WAI. Question 3, which involves the number of current diseases diagnosed by a physician, was omitted because this parameter was unlikely to reflect change due to treatment. Question 5 (sick leave during the past year) was replaced with the previous question concerning sick leave days.WAI scores range from 7 (worst) to 49 (best).
Time Frame: Baseline and 6, 12, 24, 36, 48, and 60 months
Population: Participants who were employed outside of the home, on either a part-time or full-time basis, at baseline (employed patient set) and at each time point, and with available WAI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 2110
units on a scale
  Month 6: number analyzed (Participants) | 1908
  Month 6 | 2.5 (5.9)
  Month 12: number analyzed (Participants) | 1442
  Month 12 | 3.0 (6.7)
  Month 24: number analyzed (Participants) | 986
  Month 24 | 3.2 (6.8)
  Month 36: number analyzed (Participants) | 666
  Month 36 | 3.6 (7.0)
  Month 48: number analyzed (Participants) | 452
  Month 48 | 3.3 (6.6)
  Month 60: number analyzed (Participants) | 318
  Month 60 | 3.0 (7.0)

8. Primary Outcome: Change From Baseline in Disease Activity Score - 28 Joints (DAS28)
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score < 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission.
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: Participants with sufficient data to evaluate clinical outcomes and baseline disease activity high enough to evaluate effectiveness (full analysis set), and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 4466
units on a scale
  Month 3: number analyzed (Participants) | 3749
  Month 3 | -1.34 (1.39)
  Month 6: number analyzed (Participants) | 3229
  Month 6 | -1.56 (1.46)
  Month 12: number analyzed (Participants) | 2621
  Month 12 | -1.71 (1.55)
  Month 24: number analyzed (Participants) | 1818
  Month 24 | -1.84 (1.57)
  Month 36: number analyzed (Participants) | 1250
  Month 36 | -1.94 (1.61)
  Month 48: number analyzed (Participants) | 912
  Month 48 | -2.01 (1.59)
  Month 60: number analyzed (Participants) | 650
  Month 60 | -2.15 (1.63)

9. Primary Outcome: Change From Baseline in Tender Joint Count
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Adalimumab
Number analyzed (Participants) | 4466
joints
  Month 3: number analyzed (Participants) | 4280
  Month 3 | -4.3 (6.2)
  Month 6: number analyzed (Participants) | 3657
  Month 6 | -4.9 (6.5)
  Month 12: number analyzed (Participants) | 2969
  Month 12 | -5.3 (6.7)
  Month 24: number analyzed (Participants) | 2095
  Month 24 | -5.6 (6.5)
  Month 36: number analyzed (Participants) | 1456
  Month 36 | -5.9 (6.7)
  Month 48: number analyzed (Participants) | 1040
  Month 48 | -6.1 (6.7)
  Month 60: number analyzed (Participants) | 752
  Month 60 | -6.4 (6.5)

10. Primary Outcome: Change From Baseline in Swollen Joint Count
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Adalimumab
Number analyzed (Participants) | 4466
joints
  Month 3: number analyzed (Participants) | 4280
  Month 3 | -3.2 (4.9)
  Month 6: number analyzed (Participants) | 3657
  Month 6 | -3.8 (5.2)
  Month 12: number analyzed (Participants) | 2969
  Month 12 | -4.1 (5.4)
  Month 24: number analyzed (Participants) | 2095
  Month 24 | -4.4 (5.6)
  Month 36: number analyzed (Participants) | 1456
  Month 36 | -4.8 (5.7)
  Month 48: number analyzed (Participants) | 1040
  Month 48 | -5.0 (5.7)
  Month 60: number analyzed (Participants) | 752
  Month 60 | -5.5 (6.1)

11. Primary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Adalimumab
Number analyzed (Participants) | 4466
mm/hr
  Month 3: number analyzed (Participants) | 3893
  Month 3 | -7.1 (20.5)
  Month 6: number analyzed (Participants) | 3321
  Month 6 | -7.9 (20.6)
  Month 12: number analyzed (Participants) | 2705
  Month 12 | -8.5 (21.6)
  Month 24: number analyzed (Participants) | 1891
  Month 24 | -9.0 (22.2)
  Month 36: number analyzed (Participants) | 1299
  Month 36 | -8.9 (22.1)
  Month 48: number analyzed (Participants) | 953
  Month 48 | -9.3 (22.7)
  Month 60: number analyzed (Participants) | 673
  Month 60 | -9.9 (22.5)

12. Primary Outcome: Change From Baseline in C-reactive Protein
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 4353
mg/L
  Month 3: number analyzed (Participants) | 3858
  Month 3 | -7.1 (45.2)
  Month 6: number analyzed (Participants) | 3296
  Month 6 | -7.3 (49.1)
  Month 12: number analyzed (Participants) | 2693
  Month 12 | -7.5 (59.4)
  Month 24: number analyzed (Participants) | 1918
  Month 24 | -8.0 (64.0)
  Month 36: number analyzed (Participants) | 1319
  Month 36 | -8.6 (65.9)
  Month 48: number analyzed (Participants) | 950
  Month 48 | -5.8 (47.5)
  Month 60: number analyzed (Participants) | 678
  Month 60 | -7.8 (39.3)

13. Primary Outcome: Change From Baseline in Health-Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing, eating, walking, and hygiene. Patients are asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 4449
units on a scale
  Month 3: number analyzed (Participants) | 4130
  Month 3 | -0.22 (0.51)
  Month 6: number analyzed (Participants) | 3537
  Month 6 | -0.24 (0.54)
  Month 12: number analyzed (Participants) | 2873
  Month 12 | -0.27 (0.58)
  Month 24: number analyzed (Participants) | 2014
  Month 24 | -0.28 (0.60)
  Month 36: number analyzed (Participants) | 1400
  Month 36 | -0.30 (0.62)
  Month 48: number analyzed (Participants) | 992
  Month 48 | -0.32 (0.61)
  Month 60: number analyzed (Participants) | 727
  Month 60 | -0.28 (0.63)

14. Primary Outcome: EuroQol-5 Dimensions (EQ-5D) Scores
Description: The EuroQol-5 Dimensions (EQ-5D) is a generic instrument for measuring health-related quality of life. The patient questionnaire consists of two parts. The first part includes statements for the following five areas (dimensions):
  * agility/mobility
  * self-care
  * usual activities
  * pain, bodily discomfort
  * anxiety, depression
  For each dimension the patient is asked for a three-level assessment of their health on the current day: "no problems" (1), "some problems" (2), "extreme problems" (3).
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Month 0 - at enrollment
- Month 3: 3 months after enrollment
- Month 6: 6 months after enrollment
- Month 12: 12 months after enrollment
- Month 24: 24 months after enrollment
- Month 36: 36 months after enrollment
- Month 48: 48 months after enrollment
- Month 60: 60 months after enrollment
Arm/Group | Baseline | Month 3 | Month 6 | Month 12 | Month 24 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 4400 | 4118 | 3524 | 2856 | 2020 | 1401 | 992 | 732
Participants
  Mobility: number analyzed (Participants) | 4398 | 4118 | 3524 | 2856 | 2020 | 1401 | 992 | 732
  Mobility: No problems | 1662 | 2072 | 1937 | 1644 | 1190 | 843 | 614 | 447
  Mobility: Some problems | 2728 | 2034 | 1575 | 1200 | 824 | 554 | 376 | 282
  Mobility: Extreme problems | 8 | 12 | 12 | 12 | 6 | 4 | 2 | 3
  Self-care: number analyzed (Participants) | 4394 | 4116 | 3523 | 2856 | 2020 | 1401 | 992 | 732
  Self-care: No problems | 2599 | 2792 | 2476 | 2088 | 1484 | 1038 | 729 | 506
  Self-care: Some problems | 1680 | 1226 | 972 | 706 | 503 | 338 | 243 | 208
  Self-care: Extreme problems | 115 | 98 | 75 | 62 | 33 | 25 | 20 | 18
  Usual activities: number analyzed (Participants) | 4395 | 4116 | 3523 | 2856 | 2020 | 1401 | 992 | 732
  Usual activities: No problems | 953 | 1463 | 1431 | 1303 | 958 | 677 | 503 | 353
  Usual activities: Some problems | 3236 | 2511 | 1989 | 1455 | 1015 | 696 | 464 | 362
  Usual activities: Extreme problems | 206 | 142 | 103 | 98 | 47 | 28 | 25 | 17
  Pain/discomfort: No problems | 147 | 585 | 587 | 582 | 478 | 383 | 298 | 225
  Pain/discomfort: Some problems | 2965 | 2932 | 2508 | 1989 | 1381 | 917 | 631 | 461
  Pain/discomfort: Extreme problems | 1288 | 601 | 429 | 285 | 161 | 101 | 63 | 46
  Anxiety/depression: number analyzed (Participants) | 4395 | 4116 | 3523 | 2854 | 2020 | 1400 | 992 | 732
  Anxiety/depression: No problems | 2159 | 2328 | 2141 | 1791 | 1349 | 977 | 705 | 526
  Anxiety/depression: Some problems | 1961 | 1601 | 1238 | 956 | 607 | 395 | 265 | 190
  Anxiety/depression: Extreme problems | 275 | 187 | 144 | 107 | 64 | 28 | 22 | 16

15. Primary Outcome: Change From Baseline in Euroqol Visual Analog Scale (VAS)
Description: EuroQol-5 Dimensions (EQ-5D): The EQ-5D is a generic instrument for measuring health-related quality of life. The patient questionnaire consists of two parts. The second part is a vertical, thermometer-like, VAS ranging from 0 to 100 that provides a patient-reported assessment of overall health. Patients are asked to mark how good or bad their health is on that day, with 100 meaning "the best health you can imagine" and 0 meaning "the worst health you can imagine."
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 4405
units on a scale
  Month 3: number analyzed (Participants) | 4073
  Month 3 | 10.0 (24.0)
  Month 6: number analyzed (Participants) | 3480
  Month 6 | 11.7 (24.9)
  Month 12: number analyzed (Participants) | 2815
  Month 12 | 12.9 (25.8)
  Month 24: number analyzed (Participants) | 1990
  Month 24 | 14.9 (25.4)
  Month 36: number analyzed (Participants) | 1393
  Month 36 | 16.2 (25.4)
  Month 48: number analyzed (Participants) | 986
  Month 48 | 15.8 (25.2)
  Month 60: number analyzed (Participants) | 725
  Month 60 | 14.9 (25.4)

16. Secondary Outcome: Number of Physician Visits in Past 6 Months
Description: Participants self-reported the number of physician visits they had in the past 6 months.
Time Frame: Baseline, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Baseline | Month 6 | Month 12 | Month 24 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 4344 | 3408 | 2774 | 1946 | 1357 | 960 | 703
visits
  Rheumatologist | 3.3 (3.1) | 2.5 (2.7) | 2.2 (2.0) | 1.9 (1.5) | 1.8 (1.4) | 1.9 (1.4) | 1.8 (1.6)
  General practitioner | 4.0 (4.6) | 2.9 (4.4) | 2.6 (3.2) | 2.1 (2.5) | 2.1 (3.0) | 1.9 (2.4) | 1.8 (2.5)
  Orthopedic specialist | 0.9 (2.2) | 0.6 (1.9) | 0.7 (1.6) | 0.5 (1.3) | 0.5 (1.3) | 0.5 (1.0) | 0.5 (1.9)
  Other specialists | 1.2 (2.4) | 0.9 (1.8) | 0.9 (1.8) | 0.8 (1.4) | 0.8 (1.5) | 0.8 (1.5) | 0.8 (1.5)

17. Secondary Outcome: Number of Inpatient Hospitalizations in Past 6 Months
Description: Participants self-reported the number of hospitalizations they had in the past 6 months.
Time Frame: Baseline, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Adalimumab
Number analyzed (Participants) | 4344
hospitalizations
  Baseline | 0.4 (1.5)
  Month 6: number analyzed (Participants) | 3408
  Month 6 | 0.2 (1.0)
  Month 12: number analyzed (Participants) | 2774
  Month 12 | 0.2 (1.0)
  Month 24: number analyzed (Participants) | 1946
  Month 24 | 0.1 (0.5)
  Month 36: number analyzed (Participants) | 1357
  Month 36 | 0.1 (0.4)
  Month 48: number analyzed (Participants) | 960
  Month 48 | 0.1 (0.7)
  Month 60: number analyzed (Participants) | 703
  Month 60 | 0.1 (0.4)

18. Secondary Outcome: Duration of Inpatient Hospitalizations in Past 6 Months
Description: Participants who had been hospitalized were asked how many days they were hospitalized in the past 6 months.
Time Frame: Baseline, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adalimumab
Number analyzed (Participants) | 4344
days
  Baseline | 2.3 (7.3)
  Month 6: number analyzed (Participants) | 3408
  Month 6 | 1.1 (4.4)
  Month 12: number analyzed (Participants) | 2774
  Month 12 | 1.1 (4.8)
  Month 24: number analyzed (Participants) | 1946
  Month 24 | 0.8 (3.5)
  Month 36: number analyzed (Participants) | 1357
  Month 36 | 0.7 (3.1)
  Month 48: number analyzed (Participants) | 960
  Month 48 | 0.7 (3.5)
  Month 60: number analyzed (Participants) | 703
  Month 60 | 0.5 (2.4)

19. Secondary Outcome: Number of Days With Impairment of Non-Occupational Activities in Past 6 Months
Description: Patients reported the number of days that sickness affected non-occupational activities in four categories: household, child-rearing/parenting, education, and recreational (free-time). Participants with no impairment were considered to have 0 days.
Time Frame: Baseline, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Baseline | Month 6 | Month 12 | Month 24 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 3368 | 2666 | 2199 | 1572 | 1093 | 784 | 574
days
  Household | 56.9 (64.3) | 27.7 (50.6) | 22.4 (46.1) | 20.6 (46.3) | 18.2 (43.7) | 19.2 (46.1) | 16.1 (39.8)
  Child-rearing/parenting: number analyzed (Participants) | 1220 | 1068 | 896 | 654 | 435 | 300 | 195
  Child-rearing/parenting | 15.1 (41.6) | 4.7 (23.1) | 3.1 (18.1) | 2.8 (18.4) | 1.9 (13.6) | 3.0 (19.7) | 1.6 (8.2)
  Educational: number analyzed (Participants) | 975 | 887 | 750 | 558 | 379 | 257 | 168
  Educational | 8.3 (31.6) | 2.5 (17.1) | 1.6 (13.3) | 1.1 (10.1) | 1.0 (10.1) | 0.9 (11.5) | 1.4 (12.6)
  Recreational: number analyzed (Participants) | 3101 | 2467 | 2000 | 1426 | 1016 | 728 | 532
  Recreational | 59.1 (65.6) | 28.3 (50.9) | 23.0 (47.4) | 19.5 (45.0) | 18.5 (44.9) | 19.1 (46.0) | 16.3 (41.7)

20. Secondary Outcome: Duration of Morning Stiffness
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adalimumab
Number analyzed (Participants) | 4370
minutes
  Baseline | 65.3 (72.8)
  Month 3: number analyzed (Participants) | 4222
  Month 3 | 34.6 (55.6)
  Month 6: number analyzed (Participants) | 3617
  Month 6 | 27.4 (44.3)
  Month 12: number analyzed (Participants) | 2931
  Month 12 | 24.2 (43.5)
  Month 24: number analyzed (Participants) | 2070
  Month 24 | 20.9 (39.8)
  Month 36: number analyzed (Participants) | 1439
  Month 36 | 19.0 (41.0)
  Month 48: number analyzed (Participants) | 1034
  Month 48 | 15.0 (29.8)
  Month 60: number analyzed (Participants) | 743
  Month 60 | 15.2 (32.7)

21. Secondary Outcome: Participant's Assessment of Pain
Description: Participants were asked to evaluate their level of pain in the past 7 days on a scale from 0 (no pain) to 10 (unbearable pain).
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 4455
units on a scale
  Baseline | 6.1 (2.3)
  Month 3: number analyzed (Participants) | 4178
  Month 3 | 4.4 (2.5)
  Month 6: number analyzed (Participants) | 3582
  Month 6 | 4.2 (2.5)
  Month 12: number analyzed (Participants) | 2901
  Month 12 | 3.9 (2.5)
  Month 24: number analyzed (Participants) | 2045
  Month 24 | 3.7 (2.4)
  Month 36: number analyzed (Participants) | 1415
  Month 36 | 3.5 (2.4)
  Month 48: number analyzed (Participants) | 1004
  Month 48 | 3.3 (2.4)
  Month 60: number analyzed (Participants) | 730
  Month 60 | 3.3 (2.4)

22. Secondary Outcome: Participant's Assessment of Fatigue
Description: Participants were asked to indicate how much they had suffered from abnormal exhaustion and fatigue during the past 7 days on a scale from 0 (none) to 10 (strongly).
Time Frame: Baseline and 3, 6, 12, 24, 36, 48, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 4449
units on a scale
  Baseline | 5.8 (2.7)
  Month 3: number analyzed (Participants) | 4180
  Month 3 | 4.4 (2.7)
  Month 6: number analyzed (Participants) | 3580
  Month 6 | 4.2 (2.7)
  Month 12: number analyzed (Participants) | 2901
  Month 12 | 4.0 (2.7)
  Month 24: number analyzed (Participants) | 2046
  Month 24 | 3.8 (2.7)
  Month 36: number analyzed (Participants) | 1418
  Month 36 | 3.5 (2.6)
  Month 48: number analyzed (Participants) | 1005
  Month 48 | 3.5 (2.6)
  Month 60: number analyzed (Participants) | 732
  Month 60 | 3.4 (2.7)

23. Secondary Outcome: Percentage of Participants Taking Concomitant RA Medications
Description: Assessment of concomitant medications included disease-modifying antirheumatic drugs (DMARDs) (methotrexate, Leflunomid, sulfasalazine), systemic glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), Cox-2 inhibitors (coxibs), analgesics and others.
Time Frame: Baseline to month 60
Population: Participants with sufficient data to evaluate clinical outcomes and baseline disease activity high enough to evaluate effectiveness (full analysis set).
Measure: Number; unit: percentage of participants
Groups:
- Any Visit: From baseline to month 60
Arm/Group | Baseline | Any Visit
Number analyzed (Participants) | 4466 | 4466
percentage of participants
  Methotrexate | 53.4 | 58.6
  Leflunomide | 12.0 | 13.0
  Sulfasalazine | 3.6 | 4.1
  Analgesics | 10.9 | 12.5
  NSAIDs or coxibs | 22.1 | 24.2
  Systemic glucocorticoids | 68.1 | 73.4
  Other | 3.8 | 9.8

24. Secondary Outcome: Patient Assessment of Adalimumab Therapy
Description: Participants were asked to rate therapy with adalimumab in comparison with other previous therapies according to the following response options:
  * Considerably better
  * Better
  * About the same
  * Worse
  * Noticeably worse
Time Frame: Months 3, 6, 12, 24, 36, 48, and 60
Population: Participants with sufficient data to evaluate clinical outcomes and baseline disease activity high enough to evaluate effectiveness (full analysis set), with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Month 3 | Month 6 | Month 12 | Month 24 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 4007 | 3452 | 2814 | 1983 | 1366 | 971 | 716
percentage of participants
  Considerably better | 35.6 | 39.6 | 46.3 | 51.6 | 51.5 | 55.5 | 53.6
  Better | 36.6 | 39.7 | 37.3 | 37.1 | 40.4 | 38.1 | 38.8
  About the same | 19.2 | 14.9 | 12.2 | 9.1 | 6.7 | 5.6 | 5.6
  Worse | 6.9 | 5.0 | 3.8 | 1.9 | 1.3 | 0.5 | 1.1
  Noticeably worse | 1.6 | 0.9 | 0.4 | 0.3 | 0.1 | 0.3 | 0.8

ADVERSE EVENTS:
Time Frame: 60 months
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 23/7229
Serious Adverse Events (participants affected / at risk) | 932/7229
Other Adverse Events (participants affected / at risk) | 831/7229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=7229)
Hospitalisation (Surgical and medical procedures) | 110
Knee arthroplasty (Surgical and medical procedures) | 30
Elective surgery (Surgical and medical procedures) | 27
Arthrodesis (Surgical and medical procedures) | 25
Hip arthroplasty (Surgical and medical procedures) | 24
Synovectomy (Surgical and medical procedures) | 19
Foot operation (Surgical and medical procedures) | 18
Joint arthroplasty (Surgical and medical procedures) | 18
Bunion operation (Surgical and medical procedures) | 14
Cholecystectomy (Surgical and medical procedures) | 12
Therapy cessation (Surgical and medical procedures) | 12
Surgery (Surgical and medical procedures) | 10
Therapy change (Surgical and medical procedures) | 10
Rehabilitation therapy (Surgical and medical procedures) | 9
Laparoscopic surgery (Surgical and medical procedures) | 8
Spinal operation (Surgical and medical procedures) | 8
Coronary arterial stent insertion (Surgical and medical procedures) | 7
Intervertebral disc operation (Surgical and medical procedures) | 7
Osteosynthesis (Surgical and medical procedures) | 7
Osteotomy (Surgical and medical procedures) | 7
Antibiotic therapy (Surgical and medical procedures) | 6
Arthroscopic surgery (Surgical and medical procedures) | 6
Coronary artery bypass (Surgical and medical procedures) | 6
Knee operation (Surgical and medical procedures) | 6
Rheumatoid nodule removal (Surgical and medical procedures) | 6
Antibiotic prophylaxis (Surgical and medical procedures) | 5
Aortic valve replacement (Surgical and medical procedures) | 5
Bursa removal (Surgical and medical procedures) | 5
Cardiac pacemaker insertion (Surgical and medical procedures) | 5
Inguinal hernia repair (Surgical and medical procedures) | 5
Ankle arthroplasty (Surgical and medical procedures) | 4
Baker's cyst excision (Surgical and medical procedures) | 4
Cataract operation (Surgical and medical procedures) | 4
Fracture treatment (Surgical and medical procedures) | 4
Renal stone removal (Surgical and medical procedures) | 4
Rotator cuff repair (Surgical and medical procedures) | 4
Shoulder operation (Surgical and medical procedures) | 4
Spinal fusion surgery (Surgical and medical procedures) | 4
Thyroidectomy (Surgical and medical procedures) | 4
Abdominal operation (Surgical and medical procedures) | 3
Abscess drainage (Surgical and medical procedures) | 3
Ankle operation (Surgical and medical procedures) | 3
Breast conserving surgery (Surgical and medical procedures) | 3
Cancer surgery (Surgical and medical procedures) | 3
Cardiac operation (Surgical and medical procedures) | 3
Coronary angioplasty (Surgical and medical procedures) | 3
Emergency care (Surgical and medical procedures) | 3
Gallbladder operation (Surgical and medical procedures) | 3
Haematoma evacuation (Surgical and medical procedures) | 3
Hysterectomy (Surgical and medical procedures) | 3
Joint surgery (Surgical and medical procedures) | 3
Meniscus operation (Surgical and medical procedures) | 3
Pain management (Surgical and medical procedures) | 3
Shoulder arthroplasty (Surgical and medical procedures) | 3
Sigmoidectomy (Surgical and medical procedures) | 3
Skin graft (Surgical and medical procedures) | 3
Skin neoplasm excision (Surgical and medical procedures) | 3
Spinal decompression (Surgical and medical procedures) | 3
Stent placement (Surgical and medical procedures) | 3
Tendon operation (Surgical and medical procedures) | 3
Toe operation (Surgical and medical procedures) | 3
Tooth extraction (Surgical and medical procedures) | 3
Arterial stent insertion (Surgical and medical procedures) | 2
Breast reconstruction (Surgical and medical procedures) | 2
Cardiac ablation (Surgical and medical procedures) | 2
Carpal tunnel decompression (Surgical and medical procedures) | 2
Cartilage operation (Surgical and medical procedures) | 2
Chemotherapy (Surgical and medical procedures) | 2
Gastrectomy (Surgical and medical procedures) | 2
Hernia repair (Surgical and medical procedures) | 2
Hip surgery (Surgical and medical procedures) | 2
Infiltration anaesthesia (Surgical and medical procedures) | 2
Joint dislocation reduction (Surgical and medical procedures) | 2
Massage (Surgical and medical procedures) | 2
Mastectomy (Surgical and medical procedures) | 2
Medical device removal (Surgical and medical procedures) | 2
Nasal operation (Surgical and medical procedures) | 2
Nasal polypectomy (Surgical and medical procedures) | 2
Open reduction of fracture (Surgical and medical procedures) | 2
Ovarian cystectomy (Surgical and medical procedures) | 2
Postoperative care (Surgical and medical procedures) | 2
Prostatic operation (Surgical and medical procedures) | 2
Pulmonary resection (Surgical and medical procedures) | 2
Radiotherapy (Surgical and medical procedures) | 2
Removal of internal fixation (Surgical and medical procedures) | 2
Sinus operation (Surgical and medical procedures) | 2
Tendon sheath incision (Surgical and medical procedures) | 2
Tenoplasty (Surgical and medical procedures) | 2
Thyroid operation (Surgical and medical procedures) | 2
Transurethral prostatectomy (Surgical and medical procedures) | 2
Ureteral stent insertion (Surgical and medical procedures) | 2
Wound treatment (Surgical and medical procedures) | 2
Abdominal hernia repair (Surgical and medical procedures) | 1
Adhesiolysis (Surgical and medical procedures) | 1
Adrenocortical steroid therapy (Surgical and medical procedures) | 1
Aneurysm repair (Surgical and medical procedures) | 1
Angioplasty (Surgical and medical procedures) | 1
Antiallergic therapy (Surgical and medical procedures) | 1
Anticoagulant therapy (Surgical and medical procedures) | 1
Aortic aneurysm repair (Surgical and medical procedures) | 1
Appendicectomy (Surgical and medical procedures) | 1
Arterial aneurysm repair (Surgical and medical procedures) | 1
Arterial bypass operation (Surgical and medical procedures) | 1
Arterial catheterisation (Surgical and medical procedures) | 1
Arthrotomy (Surgical and medical procedures) | 1
Bone operation (Surgical and medical procedures) | 1
Bronchial lesion excision (Surgical and medical procedures) | 1
Bursal operation (Surgical and medical procedures) | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 1
Cerebrovascular operation (Surgical and medical procedures) | 1
Chest wall operation (Surgical and medical procedures) | 1
Coronary revascularisation (Surgical and medical procedures) | 1
Cryotherapy (Surgical and medical procedures) | 1
Cyst removal (Surgical and medical procedures) | 1
Debridement (Surgical and medical procedures) | 1
Diabetes mellitus management (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Femoral hernia repair (Surgical and medical procedures) | 1
Fistula repair (Surgical and medical procedures) | 1
Fluid replacement (Surgical and medical procedures) | 1
Fracture debridement (Surgical and medical procedures) | 1
Frontal sinus operation (Surgical and medical procedures) | 1
Gastric operation (Surgical and medical procedures) | 1
Gingival operation (Surgical and medical procedures) | 1
Haemostasis (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Infusion (Surgical and medical procedures) | 1
Injection (Surgical and medical procedures) | 1
Intestinal operation (Surgical and medical procedures) | 1
Jaw operation (Surgical and medical procedures) | 1
Joint debridement (Surgical and medical procedures) | 1
Joint injection (Surgical and medical procedures) | 1
Joint stabilisation (Surgical and medical procedures) | 1
Laparotomy (Surgical and medical procedures) | 1
Leg amputation (Surgical and medical procedures) | 1
Ligament operation (Surgical and medical procedures) | 1
Limb operation (Surgical and medical procedures) | 1
Lip repair (Surgical and medical procedures) | 1
Lithotripsy (Surgical and medical procedures) | 1
Lung transplant (Surgical and medical procedures) | 1
Lymphoma operation (Surgical and medical procedures) | 1
Meniscus removal (Surgical and medical procedures) | 1
Nasal septal operation (Surgical and medical procedures) | 1
Nephrectomy (Surgical and medical procedures) | 1
Nephroplasty (Surgical and medical procedures) | 1
Nephrostomy (Surgical and medical procedures) | 1
Neurectomy (Surgical and medical procedures) | 1
Oophorectomy (Surgical and medical procedures) | 1
Ossiculoplasty (Surgical and medical procedures) | 1
Ostectomy (Surgical and medical procedures) | 1
Pancreatic operation (Surgical and medical procedures) | 1
Parotidectomy (Surgical and medical procedures) | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 1
Peritoneal lavage (Surgical and medical procedures) | 1
Pharyngeal operation (Surgical and medical procedures) | 1
Polypectomy (Surgical and medical procedures) | 1
Pyeloplasty (Surgical and medical procedures) | 1
Radical prostatectomy (Surgical and medical procedures) | 1
Radioactive iodine therapy (Surgical and medical procedures) | 1
Rectal polypectomy (Surgical and medical procedures) | 1
Renal artery stent placement (Surgical and medical procedures) | 1
Resuscitation (Surgical and medical procedures) | 1
Skin lesion removal (Surgical and medical procedures) | 1
Spinal cord operation (Surgical and medical procedures) | 1
Sternotomy (Surgical and medical procedures) | 1
Therapeutic embolisation (Surgical and medical procedures) | 1
Thrombolysis (Surgical and medical procedures) | 1
Toe amputation (Surgical and medical procedures) | 1
Tongue operation (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Tumour excision (Surgical and medical procedures) | 1
Umbilical hernia repair (Surgical and medical procedures) | 1
Unevaluable therapy (Surgical and medical procedures) | 1
Ureterectomy (Surgical and medical procedures) | 1
Ureteric operation (Surgical and medical procedures) | 1
Urinary incontinence surgery (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Venous operation (Surgical and medical procedures) | 1
Vertebral body replacement (Surgical and medical procedures) | 1
Wound closure (Surgical and medical procedures) | 1
Wound drainage (Surgical and medical procedures) | 1
Wrist surgery (Surgical and medical procedures) | 1
Pneumonia (Infections and infestations) | 59
Infection (Infections and infestations) | 14
Bronchitis (Infections and infestations) | 13
Urosepsis (Infections and infestations) | 11
Diverticulitis (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Gastroenteritis (Infections and infestations) | 8
Herpes zoster (Infections and infestations) | 8
Postoperative wound infection (Infections and infestations) | 7
Abscess limb (Infections and infestations) | 6
Post procedural infection (Infections and infestations) | 6
Sepsis (Infections and infestations) | 6
Cellulitis (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 5
Device related infection (Infections and infestations) | 4
Endocarditis (Infections and infestations) | 4
Erysipelas (Infections and infestations) | 4
Meningitis (Infections and infestations) | 4
Osteomyelitis (Infections and infestations) | 4
Subcutaneous abscess (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Abscess (Infections and infestations) | 3
Gastroenteritis norovirus (Infections and infestations) | 3
Intervertebral discitis (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Tuberculosis (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 3
Appendicitis perforated (Infections and infestations) | 2
Breast abscess (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 2
Genital herpes (Infections and infestations) | 2
Infectious colitis (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Lymph node tuberculosis (Infections and infestations) | 2
Nasal herpes (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 2
Pertussis (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Vestibular neuronitis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Abscess soft tissue (Infections and infestations) | 1
Acne pustular (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Candida pneumonia (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 1
Cholangitis infective (Infections and infestations) | 1
Chronic hepatitis C (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Emphysematous cholecystitis (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gallbladder empyema (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Herpes simplex encephalitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Infected seroma (Infections and infestations) | 1
Infection susceptibility increased (Infections and infestations) | 1
Keratouveitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Meningoencephalitis herpetic (Infections and infestations) | 1
Mycobacterium marinum infection (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia escherichia (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Pneumonia necrotising (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Poliomyelitis (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Purulence (Infections and infestations) | 1
Pyonephrosis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Septic encephalopathy (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Superinfection (Infections and infestations) | 1
Testicular abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tuberculosis gastrointestinal (Infections and infestations) | 1
Tuberculosis of genitourinary system (Infections and infestations) | 1
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Wound infection bacterial (Infections and infestations) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 35
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15
Foot deformity (Musculoskeletal and connective tissue disorders) | 14
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13
Bursitis (Musculoskeletal and connective tissue disorders) | 10
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Synovial cyst (Musculoskeletal and connective tissue disorders) | 7
Synovitis (Musculoskeletal and connective tissue disorders) | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 2
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Spinal instability (Musculoskeletal and connective tissue disorders) | 2
Ankle impingement (Musculoskeletal and connective tissue disorders) | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Bursal haematoma (Musculoskeletal and connective tissue disorders) | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Felty's syndrome (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Ligament pain (Musculoskeletal and connective tissue disorders) | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
SAPHO syndrome (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 19
Femoral neck fracture (Injury, poisoning and procedural complications) | 7
Humerus fracture (Injury, poisoning and procedural complications) | 7
Multiple fractures (Injury, poisoning and procedural complications) | 7
Tendon rupture (Injury, poisoning and procedural complications) | 7
Joint dislocation (Injury, poisoning and procedural complications) | 6
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 6
Radius fracture (Injury, poisoning and procedural complications) | 6
Ulna fracture (Injury, poisoning and procedural complications) | 6
Accident at work (Injury, poisoning and procedural complications) | 5
Foot fracture (Injury, poisoning and procedural complications) | 5
Ankle fracture (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 4
Fracture displacement (Injury, poisoning and procedural complications) | 4
Tibia fracture (Injury, poisoning and procedural complications) | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 3
Road traffic accident (Injury, poisoning and procedural complications) | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3
Accident at home (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Injury (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2
Post procedural fistula (Injury, poisoning and procedural complications) | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fractured ischium (Injury, poisoning and procedural complications) | 1
Ilium fracture (Injury, poisoning and procedural complications) | 1
Kidney rupture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Nerve injury (Injury, poisoning and procedural complications) | 1
Pancreatic duct rupture (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Stab wound (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Death (General disorders) | 16
Pyrexia (General disorders) | 14
Unevaluable event (General disorders) | 12
Complication associated with device (General disorders) | 9
Impaired healing (General disorders) | 9
Drug ineffective (General disorders) | 8
Chest pain (General disorders) | 7
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 4
Pain (General disorders) | 4
Perforated ulcer (General disorders) | 4
Peripheral swelling (General disorders) | 4
Inflammation (General disorders) | 3
No adverse event (General disorders) | 3
Asthenia (General disorders) | 2
Condition aggravated (General disorders) | 2
Cyst (General disorders) | 2
General physical health deterioration (General disorders) | 2
Swelling (General disorders) | 2
Adverse drug reaction (General disorders) | 1
Chest discomfort (General disorders) | 1
Drug interaction (General disorders) | 1
Exercise tolerance decreased (General disorders) | 1
Granuloma (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site reaction (General disorders) | 1
Injection site warmth (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Oedema peripheral (General disorders) | 1
Precancerous mucosal lesion (General disorders) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign cardiac neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease mixed cellularity stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myocardial infarction (Cardiac disorders) | 15
Coronary artery disease (Cardiac disorders) | 14
Atrial fibrillation (Cardiac disorders) | 13
Acute myocardial infarction (Cardiac disorders) | 12
Cardiac failure (Cardiac disorders) | 7
Coronary artery stenosis (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 3
Aortic valve stenosis (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Angina unstable (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 2
Sinus node dysfunction (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Adams-Stokes syndrome (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 15
Cerebral infarction (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Cerebellar infarction (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 4
Epilepsy (Nervous system disorders) | 3
Hemiparesis (Nervous system disorders) | 3
Movement disorder (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 2
Dizziness postural (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Monoparesis (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Brain stem infarction (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Complex regional pain syndrome (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Gliosis (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Orthostatic intolerance (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Post polio syndrome (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Spinal cord ischaemia (Nervous system disorders) | 1
Thalamic infarction (Nervous system disorders) | 1
Toxic encephalopathy (Nervous system disorders) | 1
Vertebral artery dissection (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Inguinal hernia (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Colitis microscopic (Gastrointestinal disorders) | 2
Diverticular perforation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Erosive duodenitis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Femoral hernia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival recession (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 1
Leukoplakia oral (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatic duct stenosis (Gastrointestinal disorders) | 1
Pancreatic mass (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Rectal polyp (Gastrointestinal disorders) | 1
Salivary gland pain (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Ulcerative gastritis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 4
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1
Arthroscopy (Investigations) | 8
Blood pressure increased (Investigations) | 6
Liver function test increased (Investigations) | 5
Bronchoscopy (Investigations) | 3
Weight decreased (Investigations) | 3
Biopsy bone marrow (Investigations) | 2
Biopsy liver (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Computerised tomogram thorax abnormal (Investigations) | 2
Double stranded DNA antibody positive (Investigations) | 2
Angiogram peripheral (Investigations) | 1
Antinuclear antibody positive (Investigations) | 1
Arteriogram coronary (Investigations) | 1
Autoantibody test (Investigations) | 1
Biopsy lymph gland (Investigations) | 1
Blood bactericidal activity (Investigations) | 1
Blood calcium (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Catheterisation cardiac (Investigations) | 1
Colonoscopy normal (Investigations) | 1
DNA antibody positive (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Emergency care examination (Investigations) | 1
Endoscopic retrograde cholangiopancreatography (Investigations) | 1
Endoscopy (Investigations) | 1
Epstein-Barr virus antibody positive (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Laparoscopy (Investigations) | 1
Mediastinoscopy (Investigations) | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1
Neurological examination (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Proteus test positive (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Transaminases abnormal (Investigations) | 1
Ultrasound abdomen abnormal (Investigations) | 1
Wound healing normal (Investigations) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 7
Urticaria (Skin and subcutaneous tissue disorders) | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Lividity (Skin and subcutaneous tissue disorders) | 1
Mucocutaneous ulceration (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 9
Haematoma (Vascular disorders) | 5
Thrombosis (Vascular disorders) | 5
Deep vein thrombosis (Vascular disorders) | 4
Peripheral arterial occlusive disease (Vascular disorders) | 4
Hypertensive crisis (Vascular disorders) | 3
Aortic aneurysm (Vascular disorders) | 2
Vasculitis (Vascular disorders) | 2
Aortic dilatation (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Lymphatic fistula (Vascular disorders) | 1
Microembolism (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 5
Nephrolithiasis (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Bladder diverticulum (Renal and urinary disorders) | 1
Bladder stenosis (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 1
Stress urinary incontinence (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary tract inflammation (Renal and urinary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 10
Cholecystitis acute (Hepatobiliary disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 4
Bile duct stone (Hepatobiliary disorders) | 3
Cholangitis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 2
Biliary cirrhosis primary (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Agranulocytosis (Blood and lymphatic system disorders) | 1
Bicytopenia (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1
Erythropenia (Blood and lymphatic system disorders) | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Depression (Psychiatric disorders) | 8
Sleep disorder (Psychiatric disorders) | 2
Stress (Psychiatric disorders) | 2
Acute stress disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Panic reaction (Psychiatric disorders) | 1
Tobacco abuse (Psychiatric disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Obesity (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5
Ovarian cyst (Reproductive system and breast disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Ovarian adhesion (Reproductive system and breast disorders) | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 1
Goitre (Endocrine disorders) | 5
Thyroid mass (Endocrine disorders) | 3
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Basedow's disease (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 2
Vertigo positional (Ear and labyrinth disorders) | 2
Otosclerosis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blepharitis (Eye disorders) | 2
Cataract (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Iritis (Eye disorders) | 1
Ophthalmic vein thrombosis (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Immunosuppression (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Device dislocation (Product Issues) | 3
Device breakage (Product Issues) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Delivery (Pregnancy, puerperium and perinatal conditions) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Alcohol use (Social circumstances) | 1
Foreign travel (Social circumstances) | 1
Postmenopause (Social circumstances) | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=7229)
Bronchitis (Infections and infestations) | 177
Nasopharyngitis (Infections and infestations) | 137
Upper respiratory tract infection (Infections and infestations) | 130
Respiratory tract infection (Infections and infestations) | 106
Infection (Infections and infestations) | 88
Herpes zoster (Infections and infestations) | 79
Influenza like illness (General disorders) | 213
Therapy cessation (Surgical and medical procedures) | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: original (2008-10-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT01076205/Prot_SAP_000.pdf
  • Study Protocol: amendment (2012-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT01076205/Prot_001.pdf